CLINICAL TRIAL: NCT03017131
Title: A Phase I Open Label Clinical Trial Evaluating the Safety and Efficacy of Adoptive Transfer of NY-ESO-1 TCR Engineered Autologous T Cells in Combination With Decitabine in Patients With Recurrent or Treatment Refractory Ovarian Cancer
Brief Title: Genetically Modified T Cells and Decitabine in Treating Patients With Recurrent or Refractory Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i 283616; NCI-2016-01477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 283616 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); P50CA159981 (NIH)
Record Dates: First submitted 2016-10-19; First posted 2017-01-11 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — aldesleukin; Cyclophosphamide; Decitabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, genetically modified T cells) (Experimental): COURSE 1: Patients receive decitabine IV daily over 1 hour on days -8 to -6, cyclophosphamide IV over 2 hours on days -4 and -3, and genetically engineered NY-ESO-1-specific T lymphocytes IV and IP on day 0. Patients also receive aldesleukin SC BID on days 1-14..
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Decitabine; Biological: Genetically Engineered NY-ESO-1-specific T Lymphocytes; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Biological: Genetically Engineered NY-ESO-1-specific T Lymphocytes — Given IV and IP
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects of genetically modified T cells and decitabine in treating patients with recurrent or refractory epithelial or non-epithelial ovarian, primary peritoneal, or fallopian tube cancer that has come back or has not responded to previous treatments. White blood cells called T cells are collected via a process called leukapheresis, genetically modified to recognize and attack tumor cells, then given back to the patient. Decitabine may induce and increase the amount of the target protein NY-ESO-1 available on the surface of tumor cells. Giving genetically modified T cells and decitabine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the autologous NY-ESO-1 redirected T cell therapy in combination with decitabine and low-dose IL-2 in patients with treatment refractory or recurrent epithelial or non-epithelial ovarian, primary peritoneal or fallopian tube carcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the persistence of genetically modified cells in the peripheral blood, and at tumor sites.

II. To examine the effect of the treatment on tumor as measured by objective tumor response and progression free survival, both assessed by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).

III. To assess the occurrence of target antigen and/or major histocompatibality complex (MHC) loss variants upon disease recurrence.

TERTIARY OBJECTIVES:

I. To evaluate the post treatment phenotype and functionality of genetically modified T cells isolated from peripheral blood and from tumor sites.

II. To assess changes in immunoscore, Tregs, Myeloid cell subsets, and antigen spreading in peripheral blood and tumor site.

III. To assess the influence of demographic and disease molecular characteristics on treatment outcomes of complete response (CR) and overall survival (OS).

OUTLINE:

COURSE 1: Patients receive decitabine IV daily over 1 hour on days -8 to Day -6, cyclophosphamide IV over 2 hours on days -4 and -3, and genetically engineered NY-ESO-1-specific T lymphocytes IV and intraperitoneally (IP) on day 0. Followed by low-dose IL-2 for 2 weeks from Day 1 to Day 14..

After completion of study treatment, patients are followed up monthly at 3-9 months, every 6 months for 4 years, and then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or refractory epithelial or non-epithelial ovarian, primary peritoneal or fallopian tube carcinoma who have received platinum containing chemotherapy and either has platinum refractory or resistant disease, or if plantinum sensitive disease, have received >= 2 lines of chemotherapy. Subjects may have received PARP inhibitators , bevacizumab or immunotherapy. Non-epithelial tumors of the ovary include sarcomas, granulosa cell tumors and malignant germ cell tumors including chiriocarcinoma
* Have been informed of other treatment options
* Must be HLA- A*02;01 positive; retesting is not required for patients who have previous documented HLA-A*02;01 positivity
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of > 4 months
* At least 4 weeks from prior chemotherapy, radiotherapy or immunotherapy, or prior investigational agents
* Must have measurable disease as defined by irRECIST
* Must have adequate venous access for apheresis; (pheresis catheter placement for cell collection is allowed)
* Women of childbearing potential in agreement to use acceptable birth control methods for the duration of the study and until persistence of the study drug is no longer detected in the peripheral blood; this may be a period of several years; methods for acceptable birth control include: condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception; it is recommended that a combination of two methods be used
* Leukocytes >= 3 x 10^9/L
* Absolute neutrophil count >= 1 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin within normal institutional limits
* Aspartate Aminotransferases (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine level = 2X< upper limit of normal (ULN): if creatinine > 2XULN, creatinine clearance must be > 60ml/min
* Patient must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients receiving any other investigational agents
* Patients with active brain metastases should be excluded from this clinical trial; patients with prior history of brain metastasis who have undergone local therapy (i.e., metastasectomy and/or radiation) and show no evidence of local recurrence or progression over the past 6 months are eligible. Brain MRI as clinically indicated only
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, decitabine or other agents used in the study
* Prior malignancy (except non melanoma skin cancer) within 3 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin 2, interferon alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to study entry

  * NOTE: recent or current use of inhaled steroids is not exclusionary; if subjects are prescribed a brief course of oral corticosteroids, the use should be limited to less than 7 days
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV) as defined below, due to the immunosuppressive effects of cyclophosphamide used and the unknown risks associated with viral replication

  * Positive serology for HIV
  * Active hepatitis B infection as determined by a positive test for hepatitis B surface antigen (Ag)
  * Active hepatitis C; patients will be screened for HCV antibody; if the HCV antibody is positive, a screening HCV ribonucleic acid (RNA) by any real time polymerase chain reaction (RT PCR) or branched deoxyribose nucleic acid (bDNA) assay must be performed at screening by a local laboratory with a Clinical Laboratory Improvement Act (CLIA) certification or its equivalent; eligibility will be determined based on a negative screening value; the test is not required if documentation of a negative result of a HCV RNA test performed within 60 days prior to screening is provided
  * Serology (CMV immunoglobulin G [IgG]) positive for active CMV
* Received any previous gene therapy using an integrating vector within 6 months
* Pregnancy or breast-feeding
* Lack of availability of a patient for immunological and clinical follow up assessment
* Evidence or history of significant cardiac disease (including evidence or history of significant cardiac disease (including myocardial infarction [MI] in the past 6 months, significant cardiac arrhythmia, stage III or IV congestive heart failure [CHF]); cardiac stress test will be done as clinically indicated; (the specific test to be chosen at the discretion of the principal investigator [PI])
* Patients with pulmonary function test abnormalities as evidenced by a forced expiratory volume in 1 second to forced vital capacity ratio measurement (FEV1/FVC) < 70% of predicted for normality will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2032-03-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events as defined by National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 28 days post infusion
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles.

SECONDARY OUTCOMES:
Appearance of target antigen/major histocompatibility complex loss variants upon disease recurrence | Up to 15 years
  Will be evaluated by quantifying expression of targeted antigens/major histocompatibility complex alleles (NY-ESO-1/human leukocyte antigen-A*02) in tumor samples obtained on disease recurrence if available, and comparing those values to the pretreatment (diagnosis) samples. NY-ESO-1 expression will be evaluated by quantitative real time polymerase chain reaction immunohistochemistry. Human leukocyte antigen-A*0201 expression on samples will be evaluated by immunohistochemistry.
Clinical response rates | Up to 15 years
  Percentage of complete and partial responses and the corresponding 95% confidence interval will be calculated.
Duration of response | Up to 15 years
  Will be observed.
Immunological parameters associated with T cell persistence, bioactivity and functionality | Up to 15 years
  Will measure the pre- and post-treatment percentage of transgenic T cells in the peripheral blood, selective migration into the tumor sites, the ex-vivo immune functionality and phenotype of these cells, the modulation of cytokine milieu in serum post treatment as compared to baseline as well as the development of an expanded patient immune response against tumor via epitope spreading.
Overall survival | Up to 15 years
  Will be observed.
Progression free survival | Up to 15 years
  The median progression free survival and the corresponding 95% confidence interval will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States